



| Use patient label Patient name: | CONSENT FORM |
|---------------------------------|--------------|
| Number: | |

## A pilot study of the use of metformin to reduce airway glucose in COPD (IRAS 19/LO/0633)

Principal investigator: Professor Sebastian Johnston Please initial 1. I confirm that I have read and understand the participant information sheet dated **Version 4, 3<sup>rd</sup> August 2022** for the above study and been given a copy to keep. I have had the opportunity to ask questions and have had these answered satisfactorily. 2. I understand that participation is voluntary, and that I am free to withdraw consent at any time, without giving any reason and without my medical care or legal rights being affected. 3. I understand that sections of any of my medical notes and data collected during the study may be looked at by responsible individuals from Imperial College, Imperial College Healthcare NHS Trust or from regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to access my records. I agree to the use of my tissue samples in this research project, as 4 described on the participant information sheet. 5. I agree to give my tissue samples as a gift to be used in any future ethicallyapproved studies. I agree to my GP being informed of my participation in the study. 6. 7. I agree to take part in this research project. Name of Participant Signature Date Name of Person taking consent Signature Date

1 copy for participant; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes.